CLINICAL TRIAL: NCT00172653
Title: Assessment of Function-Related Tests for Subjects With Stiff Shoulders: Reliability, Validity, Clinical Usefulness, and Biomechanical Analysis
Brief Title: Function-Related Tests for Subjects With Stiff Shoulders: Reliability and Validity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701216
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2005-08

CONDITIONS: Stiff Shoulder
Keywords: shoulder, reliability, validity

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: functional tasks

SUMMARY:
Background:

Shoulder-related dysfunction (SD) is a common health problem in various patient populations. SD can affect an individual's ability to function independently, consequently decreasing quality of life. A battery of simple measurable function-related tests for patients with SD is important.

Objective:

The purpose of this study is to test the reliability, validity, and potential clinical use of a battery of function-related tests in patients with SD. Additionally, the biomechanical characteristics of the battery of function-related tests will be analyzed in terms of three-dimensional shoulder complex movements and associated muscular activities.

Design:

Repeated measurements and descriptive study

Methods:

The affected arms of 60 symptomatic patients with SD will be assessed by two clinicians as well as by one clinician twice to calculate intertester and intrarater reliabilities. Assessment will include self-report measures and the battery of function-related tests (hand-in-neck, hand-to-scapula, hand-to-opposite-scapula, and modified Kibler's lateral scapular slide test). Pearson correlation or Spearman's rho correlation coefficients will be calculated and the correlation matrices will be examined for evidence of convergent and discriminative validity among pain, disability, and function-related measures in patients with SD. Principle axis factor analysis will be performed on the kinematic measurements and muscular electromyography (EMG) activities to characterize the factor loading of each task.

DETAILED DESCRIPTION:
Subjects:

Subjects with SDs will be recruited from the clinics in the department of Orthopedics and Physical Medicine and Rehabilitation at National Taiwan University Hospital (NTUH). There are about three patients with SD among 40 outpatient visits from the clinics each week. It is estimated that at least two subjects with SD per week will participate in this study. Thus, it will take six months to recruit 60 subjects with SD. All patients will be recruited and tested within a 6-month period. They will receive a written and verbal explanation of the purposes and procedures of the study. If they agree to participate they will be required to sign approved informed consent forms approved by the Human Subjects Committee of NTUH.

The inclusion criteria are adults at least 18 years old. Patients with SD will have (1) a limited ROM of a shoulder joint (ROM losses of 25% or greater compared with the noninvolved shoulder in at least two of the following shoulder motions: glenohumeral flexion, abduction, or medial/lateral rotation), and (2) pain and stiffness in the shoulder region for at least three months, and (3) the consent of the patient's physician to participate in the study. Patients with SD will be excluded after an examination by a physical therapist if they have (1) reproduction of cervical symptoms during a cervical screening examination (active and resisted range of motion, active and resisted range of motion with overpressure, quadrant test), (2) numbness or tingling in the upper extremity, (3) a history of onset of symptoms due to traumatic injury, glenohumeral or AC joint dislocation; or (4) surgery on the shoulder.

Function-related tests:

Hand-in-neck:

The hand-in-neck test will be scored on a 5-point scale, where zero represents normal function and four indicates the most decreased function (Table 1) [Mannerkorpi et al., 1999]. For this test, patients will stand and place their hands over the posterior aspect of the neck. The test performance of the patients with fibromyalgia is significantly decreased in comparison with healthy subjects [Mannerkorpi et al., 1999]. It is not known, however, to what extent performance is compromised in patients with SD.

Hand-to-scapula:

The hand-to-scapula test will be scored on a 5-point scale, where zero represents normal function and 4 indicates the most decreased function (Table 1) [Mannerkorpi et al., 1999]. This is a common task that is performed with difficulty by patients with limited range of motion of the shoulder joint. The test performance of the patients with fibromyalgia is also significantly decreased in comparison with healthy subjects [Mannerkorpi et al., 1999].

Hand-to-opposite-scapula:

The hand-to-opposite-scapula test will be scored on a 4-point scale, where zero represents normal function and three indicates the most decreased function (Table 1).

Modified Kibler's lateral scapular slide test:

Kibler et al. [1998 and 2002] characterized the scapula dysfunction by side-to-side comparisons of the scapular during arm elevation as well as at 3 test positions (Table 1). Measurements of scapula symmetry are taken bilaterally from the inferior angle of both scapulas. In this study, we will use the modified Kibler's lateral scapular slide test (LSST). The observed difference will be assessed on a three-point scale (Table. 1). The reliability and validity of the test will be assessed in patients with SD.

Pain:

Measures of pain will be included to assess validity. The patient will be asked to rate pain with movement according to a scale in which no pain will be assigned 0 points and the worst possible pain will be assigned 10 points.

Self-report measures:

Self-report measures are valuable, since they present patients' perceptions of the multifaceted effects of shoulder disorders. The literature shows that various self-report scales for the assessment of functional limitation and disability of the shoulder are available [Michener and Leggin, 2001]. Each scale is different because the developers of each questionnaire placed a particular emphasis on the selection of items from the vast range of symptoms in patients with shoulder disorders. The selection of the disabilities of the arm, shoulder and hand (DASH) and Flexilevel Scale of Shoulder Function (FLEX-SF) to assess shoulder function and disability in our study is based on its entire continuum assessment of shoulder functions and appropriate psychometric properties of reliability, validity, and responsiveness to clinical change [Beaton et al., 2001; Cook et al., 2003].

DASH:

The DASH outcome measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in subjects with any musculoskeletal disorder of the upper extremity. Beaton et al. [2001] evaluated the reliability, validity, and responsiveness of the DASH in two hundred patients with shoulder problems and demonstrated good validity, test-retest reliability, and responsiveness of the DASH. The DASH is scaled on a 0-100 score. A higher score indicates greater disability.

DASH disability/symptom score = [(sum of n responses) /n - 1] x 25 n is equal to the number of completed responses.

FLEX-SF:

In this scale, respondents answer a single question that grossly classifies their level of function as low, medium, or high. They then respond to only the items that target their level of function. Scores are recorded from 1, with the most limited function, to 50 without any limited function in the subject. This scale has been tested on 400 subjects with SDs and has showed high reliability (intraclass correlation coefficient [3,1] = 0.90) and good validity (Guyatt responsiveness index = 1.12) [Cook et al., 2003].

Quality of life:

Quality of life will be assessed on a 10-cm visual analog scale on which 0 cm indicates an excellent quality of life and 10 cm indicates the worst imaginable.

Instrumentation:

The FASTRAK motion analysis system (Polhemus Inc., Colchester, VT, USA) and a surface electromyography (sEMG) device will be used to detect shoulder complex movements and associated muscle activities. The sEMG assemblies include differential silver-silver chloride surface electrodes (an inter-electrode distance of 30 mm, 4 mm diameter), a pre-amplifier headbox (with a gain of 150), and a Bagnoli-8 amplifier (DelSys Inc., PO Box 15734, Boston, MA, USA), which has a gain of 1000, a high input impedance (10 M Ohm at 60 Hz), a common mode rejection ratio of 92 dB at 60 Hz, and a bandwidth (-3 dB) of 20 to 500 Hz. The sEMG data will be collected at 2500 Hz/channel using a 16-bit A/D board. Full bandwidth sEMG data will be reduced using a root mean square (RMS) algorithm to produce sEMG envelopes with an effective sampling rate of 20 s/s. These envelope data will be the basis for subsequent processing. Our previous investigation demonstrated that this system has good reliability to characterize functional tasks [Lin et al., 2004].

Procedures:

Reliability, validity, and potential clinical use of a battery of function-related tests:

Demographic information, physical examination, completion of pain scale report, and self-report measures (DASH and FLEX-SF) will be assessed for all patients. Two physical therapists with a minimum of 5 years' clinical experience will independently measure patients with function-related tests in each test session. One of the two testers will measure patients with function-related tests twice with 3 to 5 days' separation.

Biomechanical characteristics of the battery of function-related tests:

Surface electrodes will be placed over the upper trapezius muscle (two thirds of the distance from the spinous process of the seventh cervical vertebra to the acromion process), the lower trapezius muscle (one fourth of the distance from the thoracic spine to the inferior angle of the scapula when the arm is fully flexed in the sagittal plane), and the lower serratus anterior muscle (over the muscle fibers anterior to the latissimus dorsi muscle when the arm is flexed 90° in the sagittal plane) [Perotto, 1994]. Verification of signal quality will be investigated for each muscle by having the subject perform a resisted contraction in manual muscle test positions specific to each muscle of interest. The FASTRAK sensors will next be attached with adhesive tape to the sternum and to the skin overlying the flat superior bony surface of the scapular acromial process. A third sensor will be attached to the distal humerus between lateral and medial epicondyles with adhesive tape. These surface sensor placements are believed to have fewer skin movement artifacts. A fourth sensor will be attached to an object according to the tested functional tasks. In addition, another sensor attached to a stylus will be used to manually digitize palpated anatomical coordinates. Kinematic and EMG data will then be collected for 5 seconds in this resting seated posture. Subjects will then be asked to perform the battery of function-related tasks.

The order of function-related tasks will be randomized. Once the subjects are familiar with the functional tasks, synchronized kinematic and EMG data from 3 trials for each testing task will be collected. Subjects will be given approximately 2 to 3 minutes of rest between practice and test conditions. All subjects will be queried regarding the need for additional rest to prevent fatigue. Sensors will not be removed and replaced between trials. Data reduction will follow the method we presented in a previous published study [Lin et al., 2004].

Data analysis:

Reliability:

Descriptive statistics including means and standard deviations will be calculated for each trial and for each tester. For the intratester reliability of each measure by the same tester, data from the two test days, which will be 3 to 5 days apart, will be used to calculate kappa statistics. For the intertester reliability of each measure by the two testers, data within the test session, which will be at most 20 minutes, will be used to calculate kappa statistics.

Validity:

All the measures used in the calculation of Pearson correlation or Spearman's rho correlation coefficients will be individual trial measures. For the intratester or intertester reliability of measures (hand-to-scapula, hand-to-opposite-scapula, and modified Kibler's LSST positions 1 and 2), and the measured outcome on trial 1, tester 1 will be used. The average of the test-retest result will be used in the correlation analysis. Pearson correlation or Spearman's rho correlation coefficients will be calculated, and the correlation matrices will be examined for evidence of convergent and discriminative validity among pain, disability, and function-related measures in patients with SD.

Biomechanical characteristics of the battery of function-related tests:

Principle axis factor analysis will be performed on the kinematic measurements and muscular EMG activities to characterize the factor loading of each task. The kinematic measurements (dependent variables) will include reliable angular variable from peak scapular upward rotation, peak scapular tipping, peak scapular protraction, peak humeral elevation, peak scapular elevation, plane of humeral elevation, and humeral rotation during the testing tasks. The muscle EMG (dependent variables) will include reliable mean RMS percentages from the upper trapezius, lower trapezius, and serratus anterior during the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SD will have:

  1. A limited ROM of a shoulder joint (ROM losses of 25% or greater compared with the noninvolved shoulder in at least two of the following shoulder motions: glenohumeral flexion, abduction, or medial/lateral rotation)
  2. Pain and stiffness in the shoulder region for at least three months
  3. The consent of the patient's physician to participate in the study

Exclusion Criteria:

* Patients with SD will be excluded after an examination by a physical therapist if they have:

  1. Reproduction of cervical symptoms during a cervical screening examination (active and resisted range of motion, active and resisted range of motion with overpressure, quadrant test)
  2. Numbness or tingling in the upper extremity
  3. A history of onset of symptoms due to traumatic injury, glenohumeral or acromioclavicular (AC) joint dislocation
  4. Surgery on the shoulder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-jenq Lin, Principal Investigator — School of Physical Therapy, National Taiwan University
Locations (1):
- School of Physical Therapy, Taipei, Taiwan